CLINICAL TRIAL: NCT03008460
Title: Efficacy, Safety and Tolerability of a Bowel Cleansing Preparation (Eziclen/Izinova®) in Paediatric Subjects Undergoing Colonoscopy: a Phase III, Multicentre, Randomised, Comparative Study Versus Klean-Prep® (PEG-Electrolytes), Administered on the Day Before Colonoscopy, Investigator-blinded, Non-inferiority in Adolescents of 12 to 17 Years of Age (Inclusive) >40 kg
Brief Title: Efficacy, Safety and Tolerability of Eziclen®/Izinova® Versus Klean-prep® on Bowel Cleansing in Adolescents Undergoing Colonoscopy
Acronym: EASYKID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: F-FR-58800-003; 2016-002265-60 (EudraCT Number)
Record Dates: First submitted 2016-12-30; First posted 2017-01-02 (Estimated); Results first posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Digestive System Disease
Keywords: Bowel preparation
MeSH Terms: conditions — Digestive System Diseases | interventions — klean prep

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eziclen®/Izinova® (Experimental)
  Interventions: Drug: Eziclen®/Izinova®
- Klean-Prep® (Active Comparator)
  Interventions: Drug: Klean-Prep®

INTERVENTIONS:
Drug: Eziclen®/Izinova® — Oral solution taken the evening before the colonoscopy
  Other Names: Suprep®
  Arms: Eziclen®/Izinova®
Drug: Klean-Prep® — Oral solution taken the evening before the colonoscopy
  Arms: Klean-Prep®

SUMMARY:
The purpose of the protocol is to demonstrate that Eziclen®/Izinova®, an osmotic sulphate-based laxative preparation given on the day before colonoscopy has non-inferior efficacy to Klean-Prep® (polyethylene glycol (PEG)-electrolytes) on colon cleansing in adolescents aged 12 to 17 years (inclusive) with a body weight >40 kg, scheduled to undergo a colonoscopy for a routinely accepted diagnostic indication.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent form to participate in the study obtained from the adolescent's parent(s)/ legal representative and a signed assent form from the adolescent according to local law
* Male or female subjects between 12 to 17 years of age (inclusive)
* Body weight more than 40 kg
* Female of childbearing potential must have a negative pregnancy test
* If female, and of child-bearing potential, subject must use an acceptable form of birth control (hormonal birth control, intrauterine device (IUD), double-barrier method, or depot contraceptive)
* Routinely accepted indication for undergoing colonoscopy, including but not limited to polyposis coli diagnosis or surveillance, gastrointestinal bleeding, unexplained diarrhoea or constipation, surveillance of inflammatory bowel disease or confirmation of mucosal healing, abdominal pain, abnormal endosonography or manometry, anaemia of unknown aetiology, cancer surveillance
* In the investigator's judgment, the parent(s)/legal representative are/is mentally competent to provide informed consent for the subject to participate in the study
* In the investigator's judgement, subject is able and willing to follow study procedures including drug administration and response to questionnaires

Exclusion Criteria:

* Subject with known or suspected ileus, gastrointestinal obstruction, gastric retention (gastroparesis), rectal impaction, toxic colitis, severe ulcerative colitis or toxic megacolon, advanced carcinoma, swallowing disorders
* Subject with known or suspected inflammatory bowel disease (Crohn's disease, ulcerative colitis) in moderate to severe active phase defined by Paediatric Crohn's Disease Activity Index (PCDAI) >30 or Paediatric Ulcerative Colitis Index (PUCAI) >34
* Subject with bowel perforation or increased risk of bowel perforation, including connective tissue disorders or recent bowel surgery
* Subject with previous significant gastrointestinal surgery (e.g. colostomy, colectomy, gastric bypass, stomach stapling)
* Subject with uncontrolled pre-existing electrolyte abnormalities, or with electrolyte abnormalities based on Visit 1 laboratory results such as hypernatremia, hyponatremia, hyperphosphatemia, hypokalaemia, hypocalcaemia, uncorrected dehydration, or secondary to the use of medications such as diuretics or angiotensin converting enzyme inhibitors judged clinically significant by the investigator
* Subject with a prior history or current condition of severe renal (estimated glomerular filtration rate (GFR) less than 30 mL/min/1.73 m^2 as calculated by using the Schwartz bedside equation* [Schwartz et al, 2009]**), liver (ascites, Child-Pugh C), cardiac insufficiency (including congestive heart failure all grades) or hyperuricemia

  *The estimated GFR will be calculated in patients with elevated creatinine at baseline

  **Schwartz GJ and Work DF. Measurement and Estimation of GFR in Children and Adolescents. Clin J Am Soc Nephrol. 2009; 4: 1832-1843
* Female subject who is pregnant or lactating
* Subject who has participated in another investigational drug treatment within the last 90 days before the first study visit
* Subject with phenylketonuria
* Subject with history of asthma or hypersensitivity to any ingredient of either drug product
* Subject for whom intake of substances likely to affect gastrointestinal motility or urinary flow rate is required
* Subject with requirement to take any other oral medication within 3 hours of starting the bowel preparation, as this may impact medication absorption
* Subject with tendency for nausea and/or vomiting
* Subject with impaired consciousness that predisposes them to pulmonary aspiration or who have known swallowing disorders
* Subject with history of major medical/psychiatric conditions that, in the judgment of the investigator, would compromise safety in the study
* Subject with mental or psychiatric condition rendering the subject unable to understand the nature, scope and possible consequences of the study, and/or evidence of an uncooperative attitude
* Subject with a condition that, in the opinion of the investigator, might increase the risk to the subject or decrease the chance of obtaining satisfactory data needed to achieve the objectives of the study
* Subject who has previous enrolment in this study or concomitant enrolment in other clinical studies

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen Consumer Healthcare
Locations (24):
- Czechia (2):
  - Fakultní nemocnice Královské Vinohrady, Prague
  - Všeobecná fakultní nemocnice v Praze, Prague
- France (3):
  - Université de Picardie Jules Verne, Amiens
  - Hôpital Femme Mère-Enfant, Bron
  - Hôpital Necker Enfants Malades, Paris
- Germany (5):
  - Uniklinikum Essen, Essen
  - Evang Krankenhaus Hamm, Hamm
  - Universitätsklinikum Leipzig, Klinik und Poliklinik für Kinder- und Jugendmedizin, Leipzig
  - Klinikum Ulm, Ulm
  - HELIOS Klinikum Wuppertal, Wuppertal
- Italy (3):
  - ORN Santobono-Pausilipon Padiglione Santobono, Napoli
  - Ospedale "Spirito Santo" U.D.C., Pescara
  - Azienda Ospedaliero-Universitaria Sant'Andrea, Roma
- Netherlands (2):
  - AMC Emma kinderziekenhuis, Amsterdam
  - Maasstad ziekenhuis, Rotterdam
- Poland (9):
  - Copernicus Podmiot Leczniczy Sp. z.o.o, Gdansk
  - Samodzielny Publiczny Szpital Kliniczny Nr 6 Śląskiego, Katowice
  - Uniwersytecki Szpital Dziecięcy w Krakowie, Krakow
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Uniwersytecki Dziecięcy Szpital Kliniczny im. L. Zamenhofa w Białymstoku, Lublin
  - Uniwersytecki Szpital Dziecięcy w Lublinie, Lublin
  - Instytut "Pomnik - Centrum Zdrowia Dziecka", Warsaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 we Wrocławiu, Wroclaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Zabrze

REFERENCES:
- [Derived] Socha P, Posovszky C, Szychta M, Viscogliosi F, Martemucci L, Grzybowska-Chlebowczyk U, Perrot V, Kornowski A, Benninga MA; EASYKID Study Group. Phase III Randomized Non-Inferiority Study of OSS Versus PEG + Electrolyte Colonoscopy Preparation in Adolescents. J Pediatr Gastroenterol Nutr. 2023 May 1;76(5):652-659. doi: 10.1097/MPG.0000000000003745. Epub 2023 Feb 22. PMID 36821851

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in adolescents (aged 12 to 17 years inclusive) who were undergoing a colonoscopy for a routinely accepted diagnostic indication. Subjects were randomised 1:1 to Eziclen®/Izinova® (¾ of adult dose; 750 millilitres [mL] of preparation plus 1500 mL of water) or Klean-Prep® (70 mL/kilogram [kg]; maximum of 4000 mL). Subjects were randomised at 22 study centres in 6 countries.
Pre-assignment Details: The study consisted of a 1-day enrolment (Day 1, baseline) and investigator-blind label dosing period, a colonoscopy (Day 2) and a 30-day follow-up period (Day 32 [-5/+15, i.e. Day 27 to Day 47]). Subjects were expected to participate in the study for a minimum of 27 days and up to 47 days.
Groups:
- Eziclen®/Izinova®: Subjects received Eziclen®/Izinova® oral sulphate salt solution, administered as ¾ of the adult dose, as a 1-day regimen on the evening of the day before colonoscopy (Day 1). The 750 mL preparation was administered in 2 half doses as follows: the first half of preparation (375 mL) was drunk slowly in 30 minutes to 1 hour, followed by 750 mL of water over the next hour. Approximately 2 hours after starting the first half of preparation, the second half (375 mL) was drunk slowly in 30 minutes to 1 hour, followed by 750 mL of water over the next hour. Overall total volume (preparation + water) was 2250 mL (1125 mL per dose).
- Klean-Prep®: Subjects received Klean-Prep® oral solution, administered as a 70 mL/kg dose (calculated based on subject's weight) as a 1-day regimen on the evening of the day before colonoscopy (Day 1). The whole solution was administered in 2 half doses (1 litre per hour), with a 1-hour pause between the 2 half doses. Approximately 2 hours after starting the first half of preparation, the second half was drunk. The maximum global volume administered was 4000 mL (2000 mL per dose).
Period: Overall Study
Arm/Group | Eziclen®/Izinova® | Klean-Prep®
Started (Randomised) | 126 | 124
Completed | 119 | 110
Not Completed | 7 | 14
Not completed — Protocol deviation | 0 | 2
Not completed — Study drug not dispensed | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 5 | 6
Not completed — COVID-19 pandemic - consent withdrawn | 1 | 0
Not completed — End of study visit outside permitted time window | 0 | 1
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Population: The intention-to-treat (ITT) population included all randomised subjects who received even a partial dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Eziclen®/Izinova® | Klean-Prep® | Total
Number analyzed (Participants) | 125 | 116 | 241
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.1 (1.6) | 15.3 (1.6) | 15.2 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 47 | 107
  Male | 65 | 69 | 134
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 9 | 9 | 18
  Germany | 13 | 11 | 24
  Italy | 10 | 8 | 18
  Netherlands | 20 | 20 | 40
  Poland | 70 | 65 | 135
  Czechia | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Successful Overall Colon Preparation, Assessed With the Cleansing Score (4-point Scale)
Description: Blinded overall assessment of preparation efficacy (Cleansing Score) was determined by the colonoscopist upon completion of the examination, based on a 4-point scale as follows:
  * 4 (Excellent) = No more than small bits of adherent faeces/fluid
  * 3 (Good) = Small amounts of faeces or fluid not interfering with examination
  * 2 (Fair) = Enough faeces or fluid to prevent a completely reliable examination
  * 1 (Poor) = Large amounts of faecal residue, additional cleansing required.
  Only perfect preparations graded as excellent (4) or good (3), which allowed full, reliable examination of the mucosa were considered as successful. The adjusted percentage of subjects with a successful preparation was determined using a logistic regression model, including treatment and country as covariates.
Time Frame: At Day 2 (colonoscopy visit)
Population: The modified intention-to-treat population included all randomised subjects who received even a partial dose of study drug and produced a primary efficacy assessment.
Measure: Number (95% Confidence Interval); unit: adjusted percentage of subjects
Arm/Group | Eziclen®/Izinova® | Klean-Prep®
Number analyzed (Participants) | 125 | 116
adjusted percentage of subjects | 71.42 [56.33 to 82.89] | 79.03 [65.34 to 88.28]
Statistical Analysis 1: Comparison: Eziclen®/Izinova® vs Klean-Prep®; Analysis of the treatment difference (Eziclen®/Izinova® minus Klean-Prep®) was performed using a logistic regression model, including treatment and country as covariates; Test type: Non-Inferiority — Non-inferiority would be demonstrated if the lower limit of the 95% confidence interval of the adjusted treatment difference was higher than -15%; p = 0.0907, Regression, Logistic — P-value for non-inferiority was estimated from the adjusted treatment difference; Adjusted treatment difference = -7.61, 95% CI 2-sided [-18.45 to 3.24]

2. Secondary Outcome: Mean Colon Cleansing Score (4-point Scale)
Description: The Cleansing Score was determined by the blinded colonoscopist, based on a 4-point scale as follows:
  * 4 (Excellent) = No more than small bits of adherent faeces/fluid
  * 3 (Good) = Small amounts of faeces or fluid not interfering with examination
  * 2 (Fair) = Enough faeces or fluid to prevent a completely reliable examination
  * 1 (Poor) = Large amounts of faecal residue, additional cleansing required.
  The adjusted mean score was estimated using a 2-way analysis of variance (ANOVA), including treatment and country as covariates.
Time Frame: At Day 2 (colonoscopy visit)
Population: The ITT population included all randomised subjects who received even a partial dose of study drug.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Eziclen®/Izinova® | Klean-Prep®
Number analyzed (Participants) | 125 | 116
scores on a scale | 2.83 [2.67 to 2.99] | 3.02 [2.85 to 3.18]
Statistical Analysis 1: Comparison: Eziclen®/Izinova® vs Klean-Prep®; Analysis of the treatment difference (Eziclen®/Izinova® minus Klean-Prep®) was performed using a 2-way ANOVA, including treatment and country as covariates; Test type: Other; p = 0.0428, ANOVA; Adjusted treatment difference = -0.18, 95% CI 2-sided [-0.36 to -0.01]

3. Secondary Outcome: Mean Boston Bowel Preparation Scale (BBPS) Global Score and BBPS Scores by Colon Segment
Description: The BBPS score for each colon segment (left, transverse, right) was determined by the blinded colonoscopist as follows:
  * 0 = Unprepared colon segment with mucosa not seen due to solid stool that cannot be cleared
  * 1 = Portion of mucosa of the segment seen, but other areas of the colon segment not well seen due to staining, residual stool and/or opaque liquid
  * 2 = Minor amount of residual staining, small fragments of stool and/or opaque liquid, but mucosa of segment seen well
  * 3 = Entire mucosa of segment seen well with no residual staining, small fragments of stool and/or opaque liquid.
  Each segment score ranged from 0-3. Global score was sum of the 3 segment scores and ranged from 0-9 (worst to best). Successful colon cleansing was defined as a global BBPS score ≥6. The adjusted mean score was estimated using a 2-way ANOVA, including treatment and country as covariates.
Time Frame: At Day 2 (colonoscopy visit)
Population: The ITT population included all randomised subjects who received even a partial dose of study drug. Only subjects with data available for each specified parameter were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Eziclen®/Izinova® | Klean-Prep®
Number analyzed (Participants) | 125 | 116
scores on a scale
  Left colon: number analyzed (Participants) | 124 | 116
  Left colon | 2.05 [1.89 to 2.22] | 2.12 [1.95 to 2.29]
  Transverse colon: number analyzed (Participants) | 124 | 115
  Transverse colon | 2.25 [2.10 to 2.40] | 2.33 [2.18 to 2.48]
  Right colon: number analyzed (Participants) | 123 | 115
  Right colon | 1.92 [1.74 to 2.09] | 2.16 [1.98 to 2.34]
  Global score: number analyzed (Participants) | 123 | 115
  Global score | 6.25 [5.86 to 6.63] | 6.61 [6.21 to 7.01]
Statistical Analysis 1: Comparison: Eziclen®/Izinova® vs Klean-Prep®; Left colon: Analysis of the treatment difference (Eziclen®/Izinova® minus Klean-Prep®) was performed using a 2-way ANOVA, including treatment and country as covariates; Test type: Other; p = 0.4676, ANOVA; Adjusted treatment difference = -0.07, 95% CI 2-sided [-0.25 to 0.12]
Statistical Analysis 2: Comparison: Eziclen®/Izinova® vs Klean-Prep®; Transverse colon: Analysis of the treatment difference (Eziclen®/Izinova® minus Klean-Prep®) was performed using a 2-way ANOVA, including treatment and country as covariates; Test type: Other; p = 0.3076, ANOVA; Adjusted treatment difference = -0.09, 95% CI 2-sided [-0.25 to 0.08]
Statistical Analysis 3: Comparison: Eziclen®/Izinova® vs Klean-Prep®; Right colon: Analysis of the treatment difference (Eziclen®/Izinova® minus Klean-Prep®) was performed using a 2-way ANOVA, including treatment and country as covariates; Test type: Other; p = 0.0155, ANOVA; Adjusted treatment difference = -0.24, 95% CI 2-sided [-0.44 to -0.05]
Statistical Analysis 4: Comparison: Eziclen®/Izinova® vs Klean-Prep®; Global score: Analysis of the treatment difference (Eziclen®/Izinova® minus Klean-Prep®) was performed using a 2-way ANOVA, including treatment and country as covariates; Test type: Other; p = 0.0975, ANOVA; Adjusted treatment difference = -0.36, 95% CI 2-sided [-0.79 to 0.07]

4. Secondary Outcome: Percentage of Subjects With Need for Rescue Treatment
Description: The percentage of subjects who needed rescue treatment (saline enema) prior to colonoscopy because of inadequate preparation intake was assessed.
Time Frame: At Day 2 (colonoscopy visit, before colonoscopy)
Population: The ITT population included all randomised subjects who received even a partial dose of study drug. Only subjects with data available were included in the analysis (1 subject in the Eziclen®/Izinova® group had missing data so is not included in the overall number analysed).
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Eziclen®/Izinova® | Klean-Prep®
Number analyzed (Participants) | 124 | 116
percentage of subjects | 20.2 [13.1 to 27.2] | 14.7 [8.2 to 21.1]
Statistical Analysis 1: Comparison: Eziclen®/Izinova® vs Klean-Prep®; Analysis was performed using Cochran-Mantel-Haenszel (CMH) chi-square method (using the general association statistic), stratified on country; Test type: Other; p = 0.2428, CMH chi-square; Adjusted treatment difference rate = 1.3847, 95% CI 2-sided [0.8 to 2.4]

5. Secondary Outcome: Percentage of Subjects With Need for Nasogastric Tube To Complete Preparation
Description: The percentage of subjects who needed placement of a nasogastric tube to achieve administration of the complete preparation was assessed.
Time Frame: At Day 1 (treatment visit)
Population: The ITT population included all randomised subjects who received even a partial dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Eziclen®/Izinova® | Klean-Prep®
Number analyzed (Participants) | 125 | 116
percentage of subjects | 7.2 [2.7 to 11.7] | 31.0 [22.6 to 39.5]
Statistical Analysis 1: Comparison: Eziclen®/Izinova® vs Klean-Prep®; Analysis was performed using CMH chi-square method (using the general association statistic), stratified on country; Test type: Other; p < 0.0001, CMH chi-square; Adjusted treatment difference rate = 24.0219, 95% CI 2-sided [12.6 to 45.9]

6. Secondary Outcome: Percentage of Subjects With Colonoscopy Procedure Documented as Completed
Description: The percentage of subjects with a complete colonoscopy, defined as a procedure that reached the caecum, was assessed.
Time Frame: At Day 2 (colonoscopy visit)
Population: The ITT population included all randomised subjects who received even a partial dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Eziclen®/Izinova® | Klean-Prep®
Number analyzed (Participants) | 125 | 116
percentage of subjects | 96.8 [93.7 to 99.9] | 96.6 [93.2 to 99.9]
Statistical Analysis 1: Comparison: Eziclen®/Izinova® vs Klean-Prep®; Analysis was performed using CMH chi-square method (using the general association statistic), stratified on country; Test type: Other; p = 0.9257, CMH chi-square; Adjusted treatment difference rate = 1.0022, 95% CI 2-sided [1.0 to 1.1]

7. Secondary Outcome: Median Time to Caecal Intubation
Description: The time to caecal intubation was defined as the time from colonoscope introduction to caecal intubation, estimated using the Kaplan-Meier product limit method. In the event the procedure did not reach the caecum, the subject was censored at time of withdrawal of colonoscope.
Time Frame: From colonoscope introduction to caecal intubation, assessed on Day 2 (colonoscopy visit)
Population: The ITT population included all randomised subjects who received even a partial dose of study drug. Note: for 2 subjects in the Eziclen®/Izinova® group and 1 subject in the Klean-Prep® group, although the procedure reached the caecum, the time was not reported and consequently, these subjects could not be included in the analysis.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Eziclen®/Izinova® | Klean-Prep®
Number analyzed (Participants) | 123 | 115
minutes | 13.0 [10.0 to 15.0] | 15.0 [12.0 to 15.0]

8. Secondary Outcome: Mean Duration of Examination
Description: The duration of examination for colonoscopy (in minutes) was measured by the difference between the time of caecum intubation and the time of withdrawal of the colonoscope. The adjusted mean duration of examination was estimated using a 2-way ANOVA, including treatment and country as covariates. Subjects for whom the caecum was not reached were excluded from the analysis.
Time Frame: From caecum intubation to withdrawal of the colonoscope, assessed on Day 2 (colonoscopy visit)
Population: The ITT population included all randomised subjects who received even a partial dose of study drug. Only subjects with data available were included in the analysis (6 subjects in the Eziclen®/Izinova® group and 5 subjects in the Klean-Prep® group had missing data so are not included in the overall number analysed).
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Eziclen®/Izinova® | Klean-Prep®
Number analyzed (Participants) | 119 | 111
minutes | 14.77 [12.63 to 16.92] | 15.70 [13.50 to 17.90]
Statistical Analysis 1: Comparison: Eziclen®/Izinova® vs Klean-Prep®; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.4459, ANOVA; Adjusted treatment difference = -0.93, 95% CI 2-sided [-3.32 to 1.47]

9. Secondary Outcome: Mean Score for Overall Treatment Acceptability, Assessed Using Treatment Acceptability Questionnaire
Description: The Treatment Acceptability Questionnaire was completed by the caregiver or subject after the subject ended the intake of preparation. Subject acceptability was rated as follows:
  * 1 = Very badly accepted/unacceptable
  * 2 = Badly but accepted
  * 3 = Neither good nor bad
  * 4 = Well accepted
  * 5 = Very well accepted.
  Overall acceptability score is the average of scores from the 2 doses ranging from 1 - 5 (worst to best). The adjusted mean score was estimated using a 2-way ANOVA, including treatment and country as covariates.
Time Frame: At Day 1 (treatment visit)
Population: The ITT population included all randomised subjects who received even a partial dose of study drug. Only subjects with data available were included in the analysis (6 subjects in the Klean-Prep® group had missing data so are not included in the overall number analysed).
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Eziclen®/Izinova® | Klean-Prep®
Number analyzed (Participants) | 125 | 110
scores on a scale | 2.93 [2.65 to 3.21] | 2.22 [1.92 to 2.51]
Statistical Analysis 1: Comparison: Eziclen®/Izinova® vs Klean-Prep®; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.0001, ANOVA; Adjusted treatment difference = 0.71, 95% CI 2-sided [0.40 to 1.03]

10. Secondary Outcome: Mean Overall Treatment Compliance
Description: Treatment compliance according the instructions of use provided in the prescription was assessed as the percentage of volume of fluid taken relative to the planned volume of fluid to be taken (measured by the caregiver and reported in the treatment questionnaire of subject's leaflet during treatment administration). Overall treatment compliance was derived from the total volumes of fluid (i.e. preparation + hydration for Eziclen®/Izinova® and preparation only for Klean-Prep®) and was assessed for dose 1, dose 2 and globally (accounting for both doses). The adjusted mean overall treatment compliance (%) was estimated using a 2-way ANOVA, including treatment and country as covariates.
Time Frame: At Day 1 (treatment visit)
Population: The ITT population included all randomised subjects who received even a partial dose of study drug.
Measure: Mean (95% Confidence Interval); unit: adjusted percentage of fluid volume (mL)
Arm/Group | Eziclen®/Izinova® | Klean-Prep®
Number analyzed (Participants) | 125 | 116
adjusted percentage of fluid volume (mL)
  Dose 1 | 96.74 [94.19 to 99.30] | 95.52 [92.90 to 98.13]
  Dose 2 | 93.53 [89.24 to 97.81] | 87.14 [82.76 to 91.53]
  Global | 96.82 [93.32 to 100.31] | 89.34 [85.74 to 92.93]
Statistical Analysis 1: Comparison: Eziclen®/Izinova® vs Klean-Prep®; Dose 1: Analysis of the treatment difference (Eziclen®/Izinova® minus Klean-Prep®) was performed using a 2-way ANOVA, including treatment and country as covariates; Test type: Other; p = 0.3945, ANOVA; Adjusted treatment difference rate = 1.22, 95% CI 2-sided [-1.60 to 4.05]
Statistical Analysis 2: Comparison: Eziclen®/Izinova® vs Klean-Prep®; Dose 2: Analysis of the treatment difference (Eziclen®/Izinova® minus Klean-Prep®) was performed using a 2-way ANOVA, including treatment and country as covariates; Test type: Other; p = 0.0085, ANOVA; Adjusted treatment difference rate = 6.38, 95% CI 2-sided [1.65 to 11.12]
Statistical Analysis 3: Comparison: Eziclen®/Izinova® vs Klean-Prep®; Global: Analysis of the treatment difference (Eziclen®/Izinova® minus Klean-Prep®) was performed using a 2-way ANOVA, including treatment and country as covariates; Test type: Other; p = 0.0036, ANOVA; Adjusted treatment difference rate = 7.48, 95% CI 2-sided [2.46 to 12.50]

11. Secondary Outcome: Mean Subject Tolerability Total Score, Assessed Using a Symptom Scale
Description: Tolerability was assessed using a Symptom Scale after each dose of treatment for stomach cramping, stomach bloating and nausea on a paediatric 5-point scale as follows:
  * 1 = No symptom
  * 2 = Mild
  * 3 = Bothersome
  * 4 = Distressing
  * 5 = Severely distressing symptoms.
  The total tolerability score is the sum of the scores for the 3 symptoms ranging from 3 to 15 (best to worst). Mean total tolerability scores after dose 1 and dose 2 are presented.
Time Frame: At Day 1 (treatment visit)
Population: The safety population included all randomised subjects who received even a partial dose of study drug. Subjects were assessed according to the treatment received (1 subject randomised to the Eziclen®/Izinova® group was mistakenly administered Klean-Prep®; this subject was therefore included in the Klean-Prep® safety population).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Eziclen®/Izinova® | Klean-Prep®
Number analyzed (Participants) | 124 | 117
scores on a scale
  Dose 1 | 5.48 (2.42) | 6.34 (2.78)
  Dose 2: number analyzed (Participants) | 122 | 113
  Dose 2 | 5.93 (2.58) | 6.71 (3.07)

12. Other Pre Specified Outcome: Median Time to Clear Effluent
Description: The time to clear effluent, as reported by the subject, was defined as the time between first intake of prescription and first clear watery stool, estimated using the Kaplan-Meier product limit method. In the event of no clear watery stools, subjects with colonoscopy were censored at the time of colonoscope introduction, and subjects without colonoscopy were censored at time of start of treatment + 12 hours. Although time to clear effluent was pre-specified as a secondary endpoint in the study protocol, in a change to the planned analysis, it was subsequently analysed and reported as an 'other' efficacy endpoint.
Time Frame: From first intake of prescription to first clear watery stool, assessed on Day 1 (treatment visit) and Day 2 (colonoscopy visit)
Population: The ITT population included all randomised subjects who received even a partial dose of study drug.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Eziclen®/Izinova® | Klean-Prep®
Number analyzed (Participants) | 125 | 116
hours | 4.3 [3.5 to 5.3] | 4.8 [3.8 to 5.8]

13. Other Pre Specified Outcome: Mean Time Between Last Intake of Fluids and Start of Colonoscopy Procedure
Description: The time between the end of treatment administration (on Day 1) and the start of colonoscopy (on Day 2) was determined. The adjusted mean time between the last intake of fluids and the start of colonoscopy procedure was estimated using a 2-way ANOVA, including treatment and country as covariates.
Time Frame: From end of treatment administration to start of colonoscopy, assessed on Day 1 (treatment visit) and Day 2 (colonoscopy visit)
Population: The ITT population included all randomised subjects who received even a partial dose of study drug.
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Eziclen®/Izinova® | Klean-Prep®
Number analyzed (Participants) | 125 | 116
hours | 15.30 [14.72 to 15.88] | 14.25 [13.65 to 14.84]
Statistical Analysis 1: Comparison: Eziclen®/Izinova® vs Klean-Prep®; Analysis of the treatment difference (Eziclen®/Izinova® minus Klean-Prep®) was performed using 2-way ANOVA, including treatment and country as covariates; Test type: Other; p = 0.0015, ANOVA; Adjusted treatment difference = 1.05, 95% CI 2-sided [0.41 to 1.69]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from Day 1 up to Day 32 (30 days [-5+/15] after colonoscopy).
Description: The safety population included all randomised subjects who received even a partial dose of study drug. Subjects were assessed according to the treatment received (1 subject randomised to the Eziclen®/Izinova® group was mistakenly administered Klean-Prep®; this subject was therefore included in the Klean-Prep® safety population).
Arm/Group | Eziclen®/Izinova® | Klean-Prep®
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/117
Serious Adverse Events (participants affected / at risk) | 4/124 | 3/117
Other Adverse Events (participants affected / at risk) | 111/124 | 105/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eziclen®/Izinova® (N=124) | Klean-Prep® (N=117)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 2 (2) | 1 (1) — Diagnostic finding at colonoscopy, reported as non-related TEAE and related to the indication for colonoscopy.
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eziclen®/Izinova® (N=124) | Klean-Prep® (N=117)
Nausea (Gastrointestinal disorders) | 90 (123) | 84 (115)
Abdominal distension (Gastrointestinal disorders) | 67 (91) | 77 (107)
Abdominal pain upper (Gastrointestinal disorders) | 64 (83) | 64 (84)
Vomiting (Gastrointestinal disorders) | 11 (11) | 10 (11)
Crohn's disease (Gastrointestinal disorders) | 9 (9) | 2 (2) — Diagnostic finding at colonoscopy, reported as non-related TEAE and related to the indication for colonoscopy.
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 3 (3)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 6 (6) — Diagnostic finding at colonoscopy, reported as non-related TEAE and related to the indication for colonoscopy.
Gastritis (Gastrointestinal disorders) | 4 (4) | 3 (3)
Headache (Nervous system disorders) | 9 (9) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor requires that reasonable opportunity be given to review the content and conclusions of any abstract, presentation, or paper before the material is submitted for publication or communicated. The sponsor will comment on the draft documents within the time period agreed in the contractual arrangements. Requested amendments will be incorporated by the author, provided they do not alter the scientific value of the material.

DOCUMENTS (2):
  • Study Protocol (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/60/NCT03008460/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/60/NCT03008460/SAP_001.pdf